CLINICAL TRIAL: NCT05055908
Title: Efficacy and Biomarker Development for Lung Cancer Treated With Immune Checkpoint Inhibitors With or Without Chemotherapy
Brief Title: Efficacy and Biomarker Development for Lung Cancer Treated With Immune Checkpoint Inhibitors
Acronym: BECOME
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Hunan Province Tumor Hospital (Other)
Responsible Party: Principal Investigator, Yongchang Zhang, Professor, Director of Clinical Trial Center, Hunan Province Tumor Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20210913
Record Dates: First submitted 2021-09-15; First posted 2021-09-24 (Actual); Last update posted 2024-08-02 (Actual); Status verified 2024-07

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms | interventions — Pemetrexed; pembrolizumab; Bevacizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Cohort A: Chemotherapy plus Immune Checkpoint Inhibitors (Experimental): Lung Cancer patients treated with Chemotherapy plus Immune Checkpoint Inhibitors.
  Interventions: Drug: Pemetrexed plus Pembrolizumab
- Cohort B: Immune Checkpoint Inhibitors monotherapy (Experimental): Lung Cancer patients treated with Immune Checkpoint Inhibitors monotherapy.
  Interventions: Drug: Pembrolizumab
- Cohort C: Chemotherapy Group. (Experimental): Lung Cancer patients treated with Chemotherapy.
  Interventions: Drug: Pemetrexed

INTERVENTIONS:
Drug: Pemetrexed plus Pembrolizumab — Atezolizumab(1200mg) ivgtt, every 21 days, or pembrolizumab, 200mg ivgtt, every 21 days etc. Pemetrexed, 500mg/m2, ivgtt, every 21 days
  Other Names: Bevacizumab
  Arms: Cohort A: Chemotherapy plus Immune Checkpoint Inhibitors
Drug: Pembrolizumab — Atezolizumab(1200mg) ivgtt, every 21 days, or pembrolizumab, 200mg ivgtt, every 21 days etc.
  Arms: Cohort B: Immune Checkpoint Inhibitors monotherapy
Drug: Pemetrexed — Pemetrexed, 500mg/m2, ivgtt, every 21 days etc.
  Other Names: Bevacizumab
  Arms: Cohort C: Chemotherapy Group.

SUMMARY:
The purpose of the study is to find some biomarkers to predict the the adverse events of Immune Checkpoint Inhibitors monotherapy or plus platinum based chemotherapy in lung cancer.

DETAILED DESCRIPTION:
The purpose of the study is to find some biomarkers to predict the the adverse events of Immune Checkpoint Inhibitors monotherapy or plus platinum based chemotherapy in lung cancer.

Step 1: All the lung cancer patients treated with Immune Checkpoint Inhibitors monotherapy or plus platinum based chemotherapy were enrolled in this study.

Step 2: All the adverse events were evaluated by principal investigator. Step 3: All the blood and FFPE samples were collected for further anaysis. Step 4: Correlation between adverse events and gene profile was analysis. Step 4: Predict model was construted with AI.

ELIGIBILITY:
Inclusion Criteria:

1. Understand the requirements and contents of the clinical trial, and provide a signed and dated informed consent form.
2. Age ≥ 18 years.
3. Histologically or cytologically confirmed lung cancer.
4. Treated with Immune Checkpoint Inhibitors with or without chemotherapy.

6. Predicted survival ≥ 12 weeks. 7. Adequate bone marrow hematopoiesis and organ function 8. Presence of measurable lesions according to RECIST 1.1.

Exclusion Criteria:

Any conditions can not match for the Inclusion Criteria, includign do not have the data to perform Adverse Events evalutation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12000 (Estimated)
Dates: Start 2021-10-01 (Actual); Primary Completion 2025-07-01 (Estimated); Study Completion 2027-09-14 (Estimated)

PRIMARY OUTCOMES:
Correlation between Adverse events (AEs) and gene profile | Time from first subject dose to study completion, or up to 36 month
  Correlation between Adverse events (AEs) and gene profile

SECONDARY OUTCOMES:
Adverse events (AEs) rate according to CTCAE 5.0 | Time from first subject dose to study completion, or up to 36 month
  Adverse events (AEs) rate according to CTCAE 5.0
Correlation between Adverse events (AEs) and survival outcome | Time from first subject dose to study completion, or up to 36 month
  Correlation between Adverse events (AEs) and survival outcome

CONTACTS AND LOCATIONS:
Overall Officials: Yongchang Zhang, MD, Principal Investigator — Hunan Cancer Hospital
Locations (1):
- Hunan Cancer Hospital, Changsha, Hunan, China